CLINICAL TRIAL: NCT04371536
Title: A Single-Center, Open-Label, Randomized Feasibility Trial of Standard Oral Iron Therapy Versus Oral Iron Plus a Web-based Behavioral Intervention in Young Children With Nutritional Iron Deficiency Anemia
Brief Title: Oral Iron Versus Oral Iron Plus a Web-based Behavioral Intervention in Young Children (IRONCHILD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jacquelyn Powers, MD, MS, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-45869 IRONCHILD; K23HL132001 (NIH)
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Iron Deficiency Anemia; Iron-deficiency
Keywords: Iron Deficiency Anemia; Nutritional iron deficiency; Ferrous sulfate oral liquid formulation
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate; Iron-Dextran Complex; FIT1 protein, Arabidopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Oral iron therapy (Active Comparator): Arm A is standard oral iron therapy for 3 months.
  Interventions: Drug: Ferrous Sulfate
- Arm B: Oral iron therapy plus IRONCHILD web-based intervention (Experimental): Oral iron therapy as per Arm A plus the IRONCHILD web-based intervention aimed at promoting oral iron adherence. This web-based intervention was developed specifically for caregivers of young children with nutritional iron deficiency anemia to promote oral iron adherence.
  Interventions: Drug: Ferrous Sulfate; Behavioral: IRONCHILD

INTERVENTIONS:
Drug: Ferrous Sulfate — Patients receive ferrous sulfate 3 mg/kg elemental iron once daily in liquid formulation.
  Other Names: Feosol; Fer-Iron
Behavioral: IRONCHILD — Delivery of the intervention at each visit should take 15 minutes or less.
  * Baseline visit (Session 1) content will be viewed
  * At 1-month follow-up visit, additional (Session 2) content will be viewed
  * At 3-month final visit, patients will view final (Session 3) content
  Other Names: Web-based intervention
  Arms: Arm B: Oral iron therapy plus IRONCHILD web-based intervention

SUMMARY:
Iron deficiency anemia (IDA) affects nearly half a million young children in the United States. Most children take liquid iron medicine by mouth for at least 3 months. However, some children take longer to get better with this medicine. This study is trying to compare different ways of giving iron medicine to young children.

For young children in the US, the main cause of IDA is nutritional, or not having enough iron in the foods they eat. This often happens when kids drink too much cow milk and/or not eating enough foods that have a lot of iron. Iron deficiency is most common in children ages 1 to 4 years of age, during a time that is important for brain development. More severe and long-lasting IDA is associated with worse brain development outcomes. That is why researchers want to understand the fastest way for kids with IDA to get better.

Standard treatment is oral iron medicine for 3 to 6 months. Many children do not take their iron medicine the full amount of time needed because of side effects like abdominal discomfort, nausea, constipation, and bad taste. Different factors can contribute to patients not completing their IDA therapy. Many families do not understand how important it is to treat IDA or do not have the motivation to continue the medication.

This study will offer different methods for treating IDA, including a different method to taking the oral iron therapy.

This new method gives oral iron by increasing a family's understanding and motivation. Another research study that interviewed families of young children with IDA found ways that helped the patients to continue their therapy. Using that information, a website called IRONCHILD was created to help motivate parents to get their children to continue the oral iron medicine.

Research studies that compare these different IDA treatment methods in young children are needed and could have benefits to short-term clinical and long-term brain development. However, we do not know whether families of young children with IDA will be willing to participate in this type of study that has different treatment methods (oral iron therapy and oral iron therapy with a web-based adherence intervention).

The goal of this clinical research study is to learn which of the two methods of care will be the best way for children with iron deficiency anemia to receive therapy.

DETAILED DESCRIPTION:
First, the doctor will confirm that patients are eligible for the study. Patients will complete the following procedures:

* Medical history including prior hospitalizations, lab results, medications, diet, social and family history
* Comprehensive Physical Examination which includes measurement of vital signs, examination of the head, eyes, ears, nose, mouth, heart, lungs, abdomen, and skin.
* Blood samples: Patients will not have any extra blood draws for this study, as the investigators will draw the blood during routine blood draws. Investigators will ask to take a little extra blood (less than half a teaspoon) for research tests. All other blood draws that patients have while on study will be for routine care and not for research purposes.

Patients will be on the study for 12 weeks. Patients will receive dietary counseling on the amount of cow milk they may have and information sheets on iron-rich foods.

There are 2 different treatments in this study and patients cannot choose which treatment they receive. Instead, they will be randomly assigned to one of the two treatments. That means there is a 50-50 chance that patients will receive liquid iron medicine by itself or that patients will receive liquid iron medicine with access to the website.

Depending on which method of care patients are assigned to, they will complete the following procedures below.

1. Oral Iron Therapy:

   Patients will receive liquid iron medicine by mouth once per day for 12 weeks. Patients will first receive this medicine during their first visit.

   During the Week 4 visit, patients will compete the following procedures:
   * Blood Samples: Patients will not have any extra blood draws (pokes) for this study as blood for research will be collected during routine blood draws. About less than half a teaspoon of extra blood will be drawn for research tests. All other blood draws that patients have while on study will be for routine care and not for research purposes
   * Focused Physical Exam which includes measurement of vital signs, examination of the eyes, mouth, heart, lungs, abdomen, and skin.
   * Patients will be asked of any side effects that they may be having.

   During the Week 8 visit, patients will return to the clinic only to pick up the oral iron medicine.

   During the Week 12 visit, patients will complete the following procedures:
   * Medical history including prior hospitalizations, lab results, medications, diet, social and family history
   * Blood Samples: Patients will not have any extra blood draws (pokes) for this study as blood for research will be collected during routine blood draws. About less than half a teaspoon of extra blood will be drawn for research tests.
   * Focused Physical Exam which includes measurement of vital signs, examination of the abdomen and skin.
   * Patients will be asked of any side effects that they may be having.
2. Oral Iron Therapy and IRONCHILD:

Patients will receive liquid iron medicine by mouth once per day for 12 weeks. Patients will receive this medication during their first visit. Patients will also be given access to a website called IRONCHILD. Patients will be shown the website, including videos, at each in-clinic visit (Baseline, Week 4, and Week 12). This website was created for patients and their parent/guardian to help patients learn more about the importance of taking their oral iron therapy.

The study team will show patients how to use the website. Patients will be given a unique log-in and password with instructions on how to access the site between visits. There are 3 sessions (one per clinic visit). One session will be completed per visit, and each session should be about 15 minutes or less. Patients will also be able to access this website from home.

During the Week 4 visit, patients will compete the following procedures:

* Blood Samples: Patients will not have any extra blood draws (pokes) for this study as blood for research will be collected during routine blood draws. About less than half a teaspoon of extra blood will be drawn for research tests. All other blood draws that patients have while on study will be for routine care and not for research purposes.
* Focused Physical Exam which includes measurement of vital signs, examination of the eyes, mouth, heart, lungs, abdomen, and skin.
* Patients will be asked of any side effects that they may be having.

During the Week 8 Visit, patients will return to the clinic only to pick up their oral iron medicine.

During the Week 12 visit, patients will complete the following procedures:

* Medical history including prior hospitalizations, lab results, medications, diet, social and family history
* Blood Samples: Patients will not have any extra blood draws (pokes) for this study as blood for research will be collected during routine blood draws. About less than half a teaspoon of extra blood will be drawn for research tests. All other blood draws that patients have while on study will be for routine care and not for research purposes
* Focused Physical Exam which includes measurement of vital signs, examination of the abdomen and skin.
* Patients will be asked of any side effects that they may be having.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 12 months to less than 48 months
2. Iron deficiency anemia (IDA) confirmed by hematologic indices and iron laboratory parameters*

   * Hgb between greater than or equal to 6 g/dL AND less than or equal to 10 g/dL
   * MCV less than or equal to 70 fl
   * Ferritin less than or equal to 15 ng/mL OR TIBC greater than or equal to 425 microgram/dL *CBC indices must be performed with 7 days of study enrollment. Iron indices must be performed within 30 days of study enrollment.
3. Clinical history consistent with nutritional IDA such as prolonged breastfeeding without adequate iron supplementation or excessive milk intake (cow milk, almond milk, soy milk, goat milk or other milk, excluding breastmilk), defined as greater than or equal to 3 cups (24 ounces)per day
4. Primary language of English or Spanish
5. Access to smartphone with data plan and/or other internet access (i.e. home computer)

Exclusion Criteria:

1. Iron deficiency likely or definitely due to blood loss from the intestine or other sites.
2. Administration of a blood transfusion
3. History or evidence of intestinal malabsorption
4. History of prior intravenous iron therapy
5. Major co-morbidity such as a serious chronic medical condition unrelated to iron deficiency apparent on history, physical examination, or laboratory tests
6. Other cause of anemia (sickle cell disease, thalassemia, bone marrow failure, etc.) apparent by history, physical examination, and/or laboratory tests.
7. Inability to tolerate oral medications
8. Other medical or social factors at discretion of treating physician

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn M Powers, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: Oral Iron Therapy Plus IRONCHILD Web-based Intervention: Oral iron therapy as per Arm A plus the IRONCHILD web-based intervention aimed at promoting oral iron adherence. This web-based intervention was developed specifically for caregivers of young children with nutritional iron deficiency anemia to promote oral iron adherence.
  Ferrous Sulfate: Patients receive ferrous sulfate 3 mg/kg elemental iron once daily in liquid formulation.
  IRONCHILD: Delivery of the intervention at each visit should take 15 minutes or less.
  * Baseline visit (Session 1) content will be viewed
  * At 1-month follow-up visit, additional (Session 2) content will be viewed
  * At 3-month final visit, patients will view final (Session 3) content
Period: Overall Study
Arm/Group | Arm A: Oral Iron Therapy | Arm B: Oral Iron Therapy Plus IRONCHILD Web-based Intervention
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled in Arm B. Due to inability to enroll on the trial, it was closed early.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Oral Iron Therapy | Arm B: Oral Iron Therapy Plus IRONCHILD Web-based Intervention | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: Years] | 2 [2 to 2] |  | 2 [2 to 2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Hemoglobin [Mean (Full Range); unit: g/dL] | 7.3 [7.3 to 7.3] |  | 7.3 [7.3 to 7.3]
Ferritin [Mean (Full Range); unit: ng/mL] | 5 [5 to 5] |  | 5 [5 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Patients Enrolled
Description: We hypothesized that 50% or more of eligible patients would enroll the study.
Time Frame: Baseline
Population: No enrolled subjects were randomized to Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Oral Iron Therapy | Arm B: Oral Iron Therapy Plus IRONCHILD Web-based Intervention
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

2. Primary Outcome: Percentage of Enrolled Subjects Who Agree With Randomization
Description: We hypothesized that randomization would be feasible, defined as agreement with randomization in greater than or equal to 80% of enrolled subjects per arm.
Time Frame: Baseline
Population: No enrolled subjects were randomized to Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Oral Iron Therapy | Arm B: Oral Iron Therapy Plus IRONCHILD Web-based Intervention
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Twelve week study period
Description: Adverse events were assessed in all enrolled subjects at all research visits.
Arm/Group | Arm A: Oral Iron Therapy | Arm B: Oral Iron Therapy Plus IRONCHILD Web-based Intervention
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Oral Iron Therapy (N=1) | Arm B: Oral Iron Therapy Plus IRONCHILD Web-based Intervention (N=0)
Emesis, Constipation (Gastrointestinal disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT04371536/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT04371536/ICF_001.pdf